CLINICAL TRIAL: NCT01464060
Title: Phase 4, Prospective, Randomized Study Comparing 14-day Non-bismuth Quadruple "Hybrid" and "Concomitant" Therapies for Helicobacter Pylori Eradication in Settings With High Clarithromycin Resistance
Brief Title: 14-day Quadruple Hybrid vs. Concomitant Therapies for Helicobacter Pylori Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Infante, Javier Molina, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INHIBRICON14
Record Dates: First submitted 2011-10-25; First posted 2011-11-03 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Quadruple therapy; Clarithromycin resistance
MeSH Terms: interventions — Amoxicillin; Metronidazole; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "Hybrid" therapy (Active Comparator): Dual therapy for 7 days: 40 mg omeprazole and 1g amoxicillin every 12h. After dual therapy continue with a quadruple therapy for 7 days: 40 mg omeprazole, 1g amoxicillin, 500 mg metronidazole and 500 mg clarithromycin every 12h.
  Interventions: Drug: PPI, amoxicillin, metronidazole and clarithromycin
- "Concomitant" therapy (Experimental): Quadruple therapy for 14 days: 40 mg omeprazole, 1g amoxicillin, 500 mg metronidazole and 500 mg clarithromycin every 12h
  Interventions: Drug: PPI, amoxicillin, metronidazole and clarithromycin

INTERVENTIONS:
Drug: PPI, amoxicillin, metronidazole and clarithromycin — Dual therapy for 7 days: 40 mg omeprazole and 1g amoxicillin every 12h. After dual therapy continue with a quadruple therapy for 7 days: 40 mg omeprazole, 1g amoxicillin, 500 mg metronidazole and 500 mg clarithromycin every 12h.
  Arms: "Hybrid" therapy
Drug: PPI, amoxicillin, metronidazole and clarithromycin — Quadruple therapy for 14 days: 40 mg omeprazole, 1g amoxicillin, 500 mg metronidazole and 500 mg clarithromycin every 12h
  Arms: "Concomitant" therapy

SUMMARY:
Helicobacter pylori (H. pylori) infects approximately 50% of the adult population and is well recognized as the main cause of gastritis, peptic ulcer disease and gastric cancer. The cure of the H. pylori infection prevents recurrence of duodenal and gastric ulcer and improves dyspepsia in a significant proportion of cases, so it is cost-effective.

Eradication therapy has changed over time. Recent meta-analyses have that the current global eradication rate after standard triple therapy (STT) is less than 80%. Several European studies have found even lower eradication rates, with 35-40% of cases resulting in treatment failure, probably due to increased resistance to antibiotics in many geographical areas, principally to clarithromycin. The usually recommended pattern in the American and European (Maastricht III) consensus conferences from 2007 has traditionally been triple therapy, composed by the combination of 2 antibiotics (clarithromycin plus amoxicillin or metronidazole) and a proton pump inhibitor (PPI) for 7-14 days. However, triple therapy was discouraged in settings with high rates of clarithromycin resistance (15-20%) and, as such, new strategies in order to improve the efficacy of first-line treatments are required. Treatment failure increases antibiotic resistant strains, leads to a second treatment and a new diagnostic test to confirm eradication. Unfortunately, it remains unknown whether there is room for improvement in these geographical areas using clarithromycin-containing therapies or switching to bismuth quadruple therapy should be followed instead.

DETAILED DESCRIPTION:
Justification of the study:

Several non-bismuth quadruple clarithromycin-containing regimens have raised over the last decade aiming to substitute standard triple therapy (STT) for first-line H. pylori eradication therapy. Sequential therapy, introduced in Italy, involves a 5-day induction phase with dual therapy (a PPI every 12 hours and amoxicillin 1g every 12 hours), followed immediately by triple therapy for 5 days with a PPI every 12 hours, metronidazole 500 mg every 12 hours and clarithromycin 500 mg every 12 hours. 10-day sequential therapy proved more effectiveness than STT with excellent treatment compliance and minimal side effects. However, the efficacy of sequential therapy seems to be notably impaired by clarithromycin resistance and dual clarithromycin and metronidazole resistance, which is becoming a common scenario in developed countries.

Other interesting and resurfaced therapeutic alternative is the non-bismuth quadruple therapy (NBQT), also called "concomitant" therapy, which includes a PPI, amoxicillin, clarithromycin and a nitroimidazole, all drugs given concurrently and twice daily. It has also demonstrated its superiority over STT and it could be potential replacement for STT as first-line regimen. However, NBQT might have several advantages over sequential therapy, namely, less complexity for both the patient and the physician, twice the duration of all prescribed antibiotics, a proper validation process worldwide and a higher efficacy over sequential therapy for both clarithromycin and dual-resistant H. pylori. Finally, another recent innovation is the 14-day quadruple clarithromycin-based regimen, so-called the sequential-concomitant "hybrid" therapy, which involves PPI and amoxicillin for 7 days plus a 7-day course of NBQT. Outstanding cure rates close to 100% have been recently reported using this scheme, thereby requiring further consideration.

Therefore it is necessary to make a controlled clinical trial to directly compare NBQT "hybrid" versus "concomitant" therapy in settings with documented high clarithromycin resistance rates. In order to maximize the efficacy of eradication regimens, it would be necessary to extend duration to 14 days and using high-dose PPI (omeprazole 40 mg bid). The results of this study will conclude whether there is still room for clarithromycin-containing regimens in H. pylori eradication even in settings with high antibiotic resistance rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyspepsia or peptic gastroduodenal ulcer for whom eradication treatment is indicated.
* Requirement of confirmation of the diagnosis of H. pylori infection by at least one positive test out of the following: breath test, histology, rapid urease test or culture.

Exclusion Criteria:

* Age less than 18 years.
* Advanced chronic disease or any other pathology that prevents attending controls and follow up.
* Allergy to any of the antibiotics in the treatment.
* Previous gastric surgery
* Pregnancy and lactation.
* History of alcohol or drug abuse.
* Previous eradication treatment.
* Consumption of antibiotics or bismuth salts during the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
"Intention to treat" eradication rates | 1 year
  "Intention-to-treat" eradication of infection.

SECONDARY OUTCOMES:
" Per protocol" eradication rate | 1 year
  " Per protocol" eradication of the infection
Treatment compliance | 1 year
Number of participants with adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Javier Molina-Infante, MD, Principal Investigator — Hospital San Pedro de Alcantara, Caceres, Spain
Locations (4):
- Azienda Ospedaliera Universitaria, Napoli, Napoli, Italy
- Spain (3):
  - Hospital de Merida, Mérida, Badajoz
  - Hospital San Pedro de Alcantara, Cáceres, Caceres
  - Hospital Virgen del Puerto, Plasencia, Caceres

REFERENCES:
- [Background] Malfertheiner P, Megraud F, O'Morain C, Bazzoli F, El-Omar E, Graham D, Hunt R, Rokkas T, Vakil N, Kuipers EJ. Current concepts in the management of Helicobacter pylori infection: the Maastricht III Consensus Report. Gut. 2007 Jun;56(6):772-81. doi: 10.1136/gut.2006.101634. Epub 2006 Dec 14. PMID 17170018
- [Background] Chey WD, Wong BC; Practice Parameters Committee of the American College of Gastroenterology. American College of Gastroenterology guideline on the management of Helicobacter pylori infection. Am J Gastroenterol. 2007 Aug;102(8):1808-25. doi: 10.1111/j.1572-0241.2007.01393.x. Epub 2007 Jun 29. PMID 17608775
- [Background] Graham DY, Shiotani A. New concepts of resistance in the treatment of Helicobacter pylori infections. Nat Clin Pract Gastroenterol Hepatol. 2008 Jun;5(6):321-31. doi: 10.1038/ncpgasthep1138. Epub 2008 Apr 29. PMID 18446147
- [Background] Megraud F. H pylori antibiotic resistance: prevalence, importance, and advances in testing. Gut. 2004 Sep;53(9):1374-84. doi: 10.1136/gut.2003.022111. No abstract available. PMID 15306603
- [Background] Graham DY, Fischbach L. Helicobacter pylori treatment in the era of increasing antibiotic resistance. Gut. 2010 Aug;59(8):1143-53. doi: 10.1136/gut.2009.192757. Epub 2010 Jun 4. PMID 20525969
- [Background] Zullo A, De Francesco V, Hassan C, Morini S, Vaira D. The sequential therapy regimen for Helicobacter pylori eradication: a pooled-data analysis. Gut. 2007 Oct;56(10):1353-7. doi: 10.1136/gut.2007.125658. Epub 2007 Jun 12. PMID 17566020
- [Background] Jafri NS, Hornung CA, Howden CW. Meta-analysis: sequential therapy appears superior to standard therapy for Helicobacter pylori infection in patients naive to treatment. Ann Intern Med. 2008 Jun 17;148(12):923-31. doi: 10.7326/0003-4819-148-12-200806170-00226. Epub 2008 May 19. PMID 18490667
- [Background] Tong JL, Ran ZH, Shen J, Xiao SD. Sequential therapy vs. standard triple therapies for Helicobacter pylori infection: a meta-analysis. J Clin Pharm Ther. 2009 Feb;34(1):41-53. doi: 10.1111/j.1365-2710.2008.00969.x. PMID 19125902
- [Background] Gatta L, Vakil N, Leandro G, Di Mario F, Vaira D. Sequential therapy or triple therapy for Helicobacter pylori infection: systematic review and meta-analysis of randomized controlled trials in adults and children. Am J Gastroenterol. 2009 Dec;104(12):3069-79; quiz 1080. doi: 10.1038/ajg.2009.555. Epub 2009 Oct 20. PMID 19844205
- [Background] Gisbert JP, Calvet X, O'Connor A, Megraud F, O'Morain CA. Sequential therapy for Helicobacter pylori eradication: a critical review. J Clin Gastroenterol. 2010 May-Jun;44(5):313-25. doi: 10.1097/MCG.0b013e3181c8a1a3. PMID 20054285
- [Background] Gisbert JP, Nyssen OP, McNicholl A, et al. Meta-analysis of sequential vs. standard triple therapy for Helicobacter pylori eradication. Helicobacter 2011;16 (Suppl 1):131.
- [Background] Prieto-Jimenez CA, Cardenas VM, Fischbach LA, Mulla ZD, Rivera JO, Dominguez DC, Graham DY, Ortiz M. Double-blind randomized trial of quadruple sequential Helicobacter pylori eradication therapy in asymptomatic infected children in El Paso, Texas. J Pediatr Gastroenterol Nutr. 2011 Mar;52(3):319-25. doi: 10.1097/MPG.0b013e318206870e. PMID 21336156
- [Background] Bontems P, Kalach N, Oderda G, Salame A, Muyshont L, Miendje DY, Raymond J, Cadranel S, Scaillon M. Sequential therapy versus tailored triple therapies for Helicobacter pylori infection in children. J Pediatr Gastroenterol Nutr. 2011 Dec;53(6):646-50. doi: 10.1097/MPG.0b013e318229c769. PMID 21701406
- [Background] Molina-Infante J, Perez-Gallardo B, Fernandez-Bermejo M, Hernandez-Alonso M, Vinagre G, Duenas C, Mateos-Rodriguez JM, Gonzalez-Garcia G, Abadia EG, Gisbert JP. Clinical trial: clarithromycin vs. levofloxacin in first-line triple and sequential regimens for Helicobacter pylori eradication. Aliment Pharmacol Ther. 2010 May;31(10):1077-84. doi: 10.1111/j.1365-2036.2010.04274.x. Epub 2010 Feb 20. PMID 20180787
- [Background] Choi WH, Park DI, Oh SJ, Baek YH, Hong CH, Hong EJ, Song MJ, Park SK, Park JH, Kim HJ, Cho YK, Sohn CI, Jeon WK, Kim BI. [Effectiveness of 10 day-sequential therapy for Helicobacter pylori eradication in Korea]. Korean J Gastroenterol. 2008 May;51(5):280-4. Korean. PMID 18516011
- [Background] Remes-Troche JM, Alarcon-Rivera G, Ramos-de la Medina A, et al. Sequential therapy vs standard triple therapy as treatment of Helicobacter pylori infection. A prospective, randomized, parallel-group, open-label study in Mexico. Gastroenterology 2010;138:S-336.
- [Background] Romano M, Cuomo A, Gravina AG, Miranda A, Iovene MR, Tiso A, Sica M, Rocco A, Salerno R, Marmo R, Federico A, Nardone G. Empirical levofloxacin-containing versus clarithromycin-containing sequential therapy for Helicobacter pylori eradication: a randomised trial. Gut. 2010 Nov;59(11):1465-70. doi: 10.1136/gut.2010.215350. PMID 20947881
- [Background] Wu DC, Hsu PI, Wu JY, Opekun AR, Kuo CH, Wu IC, Wang SS, Chen A, Hung WC, Graham DY. Sequential and concomitant therapy with four drugs is equally effective for eradication of H pylori infection. Clin Gastroenterol Hepatol. 2010 Jan;8(1):36-41.e1. doi: 10.1016/j.cgh.2009.09.030. Epub 2009 Oct 3. PMID 19804842
- [Background] Sirimontaporn N, Thong-Ngam D, Tumwasorn S, Mahachai V. Ten-day sequential therapy of Helicobacter pylori infection in Thailand. Am J Gastroenterol. 2010 May;105(5):1071-5. doi: 10.1038/ajg.2009.708. Epub 2009 Dec 15. PMID 20010919
- [Background] Mahachai V, Sirimontaporn N, Tumwasorn S, Thong-Ngam D, Vilaichone RK. Sequential therapy in clarithromycin-sensitive and -resistant Helicobacter pylori based on polymerase chain reaction molecular test. J Gastroenterol Hepatol. 2011 May;26(5):825-8. doi: 10.1111/j.1440-1746.2011.06660.x. PMID 21251064
- [Background] Vaira D, Zullo A, Vakil N, Gatta L, Ricci C, Perna F, Hassan C, Bernabucci V, Tampieri A, Morini S. Sequential therapy versus standard triple-drug therapy for Helicobacter pylori eradication: a randomized trial. Ann Intern Med. 2007 Apr 17;146(8):556-63. doi: 10.7326/0003-4819-146-8-200704170-00006. PMID 17438314
- [Background] Gisbert JP, Calvet X. Review article: non-bismuth quadruple (concomitant) therapy for eradication of Helicobater pylori. Aliment Pharmacol Ther. 2011 Sep;34(6):604-17. doi: 10.1111/j.1365-2036.2011.04770.x. Epub 2011 Jul 11. PMID 21745241
- [Background] Molina-Infante J, Pazos-Pacheco MC, Perez-Gallardo B, et al. Efficacy of non-bismuth quadruple "concomitant" therapy for H. pylori infection in a setting with high clarithromycin resistance. Gastroenterology 2011; Suppl 1:S-880.
- [Background] Hsu PI, Wu DC, Wu JY, Graham DY. Modified sequential Helicobacter pylori therapy: proton pump inhibitor and amoxicillin for 14 days with clarithromycin and metronidazole added as a quadruple (hybrid) therapy for the final 7 days. Helicobacter. 2011 Apr;16(2):139-45. doi: 10.1111/j.1523-5378.2011.00828.x. PMID 21435092
- [Background] Malfertheiner P, Bazzoli F, Delchier JC, Celinski K, Giguere M, Riviere M, Megraud F; Pylera Study Group. Helicobacter pylori eradication with a capsule containing bismuth subcitrate potassium, metronidazole, and tetracycline given with omeprazole versus clarithromycin-based triple therapy: a randomised, open-label, non-inferiority, phase 3 trial. Lancet. 2011 Mar 12;377(9769):905-13. doi: 10.1016/S0140-6736(11)60020-2. Epub 2011 Feb 21. PMID 21345487
- [Background] Dore MP, Farina V, Cuccu M, Mameli L, Massarelli G, Graham DY. Twice-a-day bismuth-containing quadruple therapy for Helicobacter pylori eradication: a randomized trial of 10 and 14 days. Helicobacter. 2011 Aug;16(4):295-300. doi: 10.1111/j.1523-5378.2011.00857.x. PMID 21762269
- [Background] Villoria A, Garcia P, Calvet X, Gisbert JP, Vergara M. Meta-analysis: high-dose proton pump inhibitors vs. standard dose in triple therapy for Helicobacter pylori eradication. Aliment Pharmacol Ther. 2008 Oct 1;28(7):868-77. doi: 10.1111/j.1365-2036.2008.03807.x. Epub 2008 Jul 17. PMID 18644011
- [Derived] Molina-Infante J, Romano M, Fernandez-Bermejo M, Federico A, Gravina AG, Pozzati L, Garcia-Abadia E, Vinagre-Rodriguez G, Martinez-Alcala C, Hernandez-Alonso M, Miranda A, Iovene MR, Pazos-Pacheco C, Gisbert JP. Optimized nonbismuth quadruple therapies cure most patients with Helicobacter pylori infection in populations with high rates of antibiotic resistance. Gastroenterology. 2013 Jul;145(1):121-128.e1. doi: 10.1053/j.gastro.2013.03.050. Epub 2013 Apr 3. PMID 23562754